CLINICAL TRIAL: NCT04542694
Title: Open-label Randomized Multicenter Comparative Study on the Efficacy and Safety of Areplivir Film-coated Tablets (PROMOMED RUS LLC, Russia) in Patients Hospitalized With COVID-19
Brief Title: Study of Favipiravir Compared to Standard of Care in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAV052020
Record Dates: First submitted 2020-09-04; First posted 2020-09-09 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
Keywords: Favipiravir; Areplivir; COVID-19; SARS-CoV-2; 2019-nCoV
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Areplivir) (Experimental): Arm 1 (n=100) receives the study drug Areplivir film-coated tablets:
  on day 1 of therapy - 1600 mg (8 tablets) 2 times a day; on days 2-14 of treatment - 600 mg (3 tablets) 2 times a day. The drug is taken orally every 12 hours, swallowing whole tablet without chewing and washing down with a glass of water. The course of treatment is 14 days. The test drug is administered in hospital setting under supervision of a clinical investigator. The test drug is not handed over to the patient.
  Interventions: Drug: Favipiravir
- Standard of care (Active Comparator): Arm 2 (n=100) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the Interim Guidelines for the prevention, diagnosis and treatment of new coronavirus infection (COVID-19) approved by the Russian Ministry of Health (but not Favipiravir) by decision of the investigator and taking into account the availability of drugs at the study site. Might include hydroxychloroquine (with or without azithromycin), chloroquine, lopinavir/ritonavir or other recommended schemes.
  Standard therapy is administered in hospital setting. Discharge of patients from a hospital is carried out in accordance with the local practice of the study site in compliance with the current sanitary and epidemiological regime.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Favipiravir — 200 mg coated tablets
  Other Names: AREPLIVIR
  Arms: Favipiravir (Areplivir)
Drug: Standard of care — Drug: Standard of Care Standard of Care will be prescribed in accordance with the recommended treatment regimens presented in the Russian guidelines for the prevention, diagnosis and treatment of COVID-19 according to the decision of the Investigator.
  Other Name: Hydroxychloroquine, chloroquine, lopinavir/ritonavir, etc.
  Arms: Standard of care

SUMMARY:
This is open-labe randomized multicenter comparative Phase III study conducted in 5 medical facilities. The objective of the study is to assess the efficacy and safety of Favipiravir compared with the Standard of care (SOC) in hospitalized patients with moderate COVID-19 pneumonia.

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 200 eligible patients with polymerase chain reaction (PCR) confirmed COVID-19 are randomized at a 1:1 ratio to receive either Favipiravir 1600 mg twice a day (BID) on Day 1 followed by 600 mg BID on Days 2-14 (1600/600 mg), or SOC. The course of treatment by Favipiravir is 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signing and dating of the Informed Consent Form of the Patient Information Leaflet (PIL) by patients.
2. Men and women aged 18 to 80 years inclusive at the time of signing the Informed Consent Form in PIL.
3. No difficulty with oral medication (e.g. swallowing disorder).
4. Patient diagnosed with "Coronavirus infection caused by SARS-CoV-2 (confirmed)1, moderate severity form*" established in accordance with the Interim Guidelines of the Russian Ministry of Health for the prevention, diagnosis and treatment of a new coronavirus infection (COVID-19), (revision 6 of 28.04.2020).

   *Moderate severity form: fever above 38 °C, BR above 22/min, dyspnea during exercise, pneumonia (confirmed by lung CT), SpO2 < 95%, C reactive protein (CRP) serum level above 10 mg/l.
5. Patient should be hospitalized no more than 48 hours before the start of the study therapy.
6. Positive PCR result for presence of SARS-CoV-2 RNA at screening phase (results obtained within 7 days prior to screening are appropriate).
7. Patient's consent to use reliable contraceptive methods throughout the study and within 1 month for women and 3 months for men after its completion. Persons eligible for participation in the study: - Women who have a negative pregnancy test and use the following contraceptives: barrier method (condom or occlusive cap (diaphragm or cervical/vaulted cap)) or double barrier method of contraception (condom or occlusive cap (diaphragm or cervical/vaulted cap) plus spermicide (foam/gel/film/cream/suppository)). Women incapable of childbearing may also participate in the study (with past history of: hysterectomy, tubal ligation, infertility, menopause more than 1 year) or men with preserved reproductive function who use barrier contraceptives, as well as men with infertility or vasectomy in the past medical history.

Exclusion Criteria:

1. Hypersensitivity to favipiravir and/or other components of the study drug.
2. Impossibility of CT procedure (for example, gypsum dressing or metal structures in the field of imaging).
3. The need to use drugs from the list of prohibited therapy.
4. Need for treatment in the intensive care unit.
5. Impaired liver function (AST and/or ALT ≥ 2 UNL and/or total bilirubin ≥ 1.5 UNL) at the time of screening.
6. Impaired kidney function (creatinine clearance according to Cockcroft-Gault formula less than 45 ml/min) at the time of screening.
7. Positive testing for HIV, syphilis, hepatitis B and/or C.
8. Chronic heart failure FC III-IV according to New York Heart Association (NYHA) functional classification.
9. Malabsorption syndrome or other clinically significant gastrointestinal disease that may affect absorption of the study drug (non-correctable vomiting, diarrhea, ulcerative colitis, and others).
10. Malignancies in the past medical history.
11. Alcohol, pharmacological and/or drug addiction in the past medical history and/or at the time of screening.
12. Schizophrenia, schizoaffective disorder, bipolar disorder, or other history of mental pathology or suspicion of their presence at the time of screening.
13. Severe, decompensated or unstable somatic diseases (any disease or condition that threaten the patient's life or impair the patient's prognosis, and also make it impossible for him/her to participate in the clinical study).
14. Any history data that the investigating physician believes could lead to complication in the interpretation of the study results or create an additional risk to the patient as a result of his/her participation in the study.
15. Patient's unwillingness or inability to comply with procedures of the Study Protocol (in the opinion of physician investigator).
16. Pregnant or nursing women or women planning pregnancy.
17. Participation in another clinical study for 3 months prior to inclusion in the study.
18. Other conditions that, according to the physician investigator, prevent the patient from being included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Pushkar, Principal Investigator — Moscow State Clinical Hospital №50
Locations (5):
- Russia (5):
  - State Clinical Hospital №50, Moscow
  - Regional Clinic Hospital of Ryazan, Ryazan
  - City Hospital N40 of Kurortny District, Saint Petersburg
  - Medical institute Ogarev Mordovia State university, Saransk
  - Smolensk clinical hospital №1, Smolensk

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study will randomize 200 patients. Given the possible non-inclusion of patients at the screening stage, the maximum number of patients to sign the Informed Consent Form in the Patient Information Leaflet and to participate in screening can be no more than 210 people.
Groups:
- Favipiravir (Areplivir): Arm 1 (n=100) receives the study drug Areplivir film-coated tablets:
  on day 1 of therapy - 1600 mg (8 tablets) 2 times a day; on days 2-14 of treatment - 600 mg (3 tablets) 2 times a day. The drug is taken orally every 12 hours, swallowing whole tablet without chewing and washing down with a glass of water. The course of treatment is 14 days. The test drug is administered in hospital setting under supervision of a clinical investigator. The test drug is not handed over to the patient.
  Favipiravir: 200 mg coated tablets
Period: Overall Study
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Started | 100 | 100
Completed | 96 | 100
Not Completed | 4 | 0
Not completed — The need for prohibited therapy | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Arm 2 (n=100) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the Interim Guidelines for the prevention, diagnosis and treatment of new coronavirus infection (COVID-19) approved by the Russian Ministry of Health (but not Favipiravir) by decision of the investigator and taking into account the availability of drugs at the study site. Might include hydroxychloroquine (with or without azithromycin), chloroquine, lopinavir/ritonavir or other recommended schemes.
  Standard therapy is administered in hospital setting. Discharge of patients from a hospital is carried out in accordance with the local practice of the study site in compliance with the current sanitary and epidemiological regime.
  Standard of care: Drug: Standard of Care Standard of Care will be prescribed in accordance with the recommended treatment regimens presented in the Russian guidelines for the prevention, diagnosis and treatment of COVID-19 according to the decision of the Investigator.
  Other Name: Hydroxychloroquine, chloroquine, lopinavir/ritonavir, etc.
- Total: Total of all reporting groups
Arm/Group | Favipiravir (Areplivir) | Standard of Care | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.38 (13.18) | 49.98 (13.06) | 49.68 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 51 | 46 | 97
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Rate of Clinical Status Improvement
Description: Rate of clinical status improvement by categorical ordinal scale of clinical status improvement by 2 or more categories by Day 10 WHO Ordinal Scale for Clinical Improvement (WHO-OSCI), 0 - uninfected (There are no clinical and virological signs of infection), 8 - dead, higher scores mean a worse outcome
Time Frame: By Visit 3, approximately 10 days
Population: Intent-tо-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 27 | 15
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; A comparative analysis of the rate of clinical status improvement by 2 or more categories. The difference in percentages between the AREPLIVIR arm and the standard therapy arm (pa-pb); Test type: Superiority; p = 0.0372, Chi-squared; The difference in proportions = 0.1313, 95% CI 2-sided [-0.0004 to 0.2367]

2. Primary Outcome: Time to Clinical Improvement
Description: Time (in days) to improvement in clinical status by WHO categorical ordinal scale of clinical status improvement.
Time Frame: 28 days
Population: patients who received at least one dose of the drug in the study and for whom there is data for at least one visit after the baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
days | 8 [6 to 10] | 12 [7 to 12]
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; Comparative analysis of time to clinical status improvement by categorical ordinal clinical improvement scale between the AREPLIVIR arm and the standard therapy arm; Test type: Superiority; p < 0.0001, Log Rank; The difference in days = 4

3. Secondary Outcome: Rate of Viral Elimination by Day 10
Description: Percentage of patients with elimination (clearance) of COVID-19 according to PCR data by day 10 (negative PCR results).
Time Frame: 10 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 98 | 79
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; Test type: Superiority; p = 0.00016, Chi-squared; The difference in percentages = 22.5

4. Secondary Outcome: Time Before the End of Fever
Description: Time (in days) before the end of fever (body temperature < 37.2 ° C for 3 consecutive days without antipyretic medication).
Time Frame: 28 days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
days | 4 [2 to 5] | 5 [3 to 7]
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; Test type: Superiority; p = 0.052, Log Rank; Median Difference (Final Values) = 1.55

5. Secondary Outcome: Change in the Level of Lung Damage According to CT
Description: Assessment of lung injury (degree of damage by "empirical" visual scale and % of patients) according to CT data comparing to baseline. The number of patients in whom by the end of therapy there was an improvement in the condition of the lungs (a decrease in the volume of the lesion according to CT)
Time Frame: Days 15, 21, 28
Population: The number of patients in whom by the end of therapy there was an improvement in the condition of the lungs (a decrease in the volume of the lesion according to CT)
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 60 | 40
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; Test type: Superiority; p = 0.1953, Chi-squared

6. Secondary Outcome: Rate of Transfer to the Intensive Care Unit
Description: Percentage of patients transferred to intensive care unit (% of patients).
Time Frame: 28 Days
Population: the number of patients who required transfer to the intensive care unit
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0
Statistical Analysis 1: Comparison: Favipiravir (Areplivir) vs Standard of Care; Test type: Superiority; p = 0.4975, Chi-squared

7. Secondary Outcome: Rate of the Use of Non-invasive Lung Ventilation
Description: Percentage of cases with non-invasive lung ventilation (% of patients).
Time Frame: 28 Days
Population: the number of patients who required non-invasive lung ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0

8. Secondary Outcome: Rate of the Use of Mechanical Ventilation
Description: Percentage of cases with mechanical lung ventilation (% of patients)
Time Frame: 28 Days
Population: the number of patients who required mechanical lung ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0

9. Secondary Outcome: Mortality
Description: Incidence of fatal cases (% of patients)
Time Frame: 28 Days
Population: the number of patients who died
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0

10. Post Hoc Outcome: Amount of Patients Without Any Clinical Signs of Disease by the Completion of Therapy (Category 0 According to a WHO Categorical Ordinal Scale)
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 44 | 10

11. Post Hoc Outcome: The Number of Patients Achieved a Category Lower Than or Equal to 2 on the WHO Clinical Improvement Scale (They Were Discharged From Hospital)
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 90 | 67

12. Post Hoc Outcome: A Number of Patients With Fever Reduction Below 37.2 ° C by the 3rd Day of Therapy
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Favipiravir (Areplivir) | Standard of Care
Number analyzed (Participants) | 100 | 100
Participants | 60 | 37

ADVERSE EVENTS:
Time Frame: Safety assessment was carried out: up to 30 days for each patient and during the entire period of the study as a whole. Safety population: patients who have received at least one dose of the study drug and for whom there is an assessment of condition and/or AE for at least one time point after administration.
Arm/Group | Favipiravir (Areplivir) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 3/100 | 0/100
Other Adverse Events (participants affected / at risk) | 25/100 | 28/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir (Areplivir) (N=100) | Standard of Care (N=100)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — According to investigators, the causal relationship with the study drug was estimated as "unrelated", SAE was associated with the presence of concomitant diseases, i.e. type 2 diabetes mellitus, obesity, and hyperthyroidism.
Multiple organ failure syndrome (General disorders) | 1 | 0 — According to investigators, the causal relationship with the study drug was estimated as "unrelated", SAE was associated with the presence of concomitant diseases, i.e. type 2 diabetes mellitus, obesity, and hyperthyroidism.
Aortic valve stenosis (Cardiac disorders) | 1 | 0 — According to investigators, the causal relationship with the study drug was estimated as "doubtful", SAE was associated with the presence of concomitant diseases, i.e. type 2 diabetes mellitus, obesity, and hyperthyroidism.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Favipiravir (Areplivir) (N=100) | Standard of Care (N=100)
Increased alanine aminotransferase activity (Hepatobiliary disorders) | 18 | 19 — According to investigators, the causal relationship with the study drug was estimated as "unrelated" in 22.2%
Increased aspartate aminotransferase activity (Hepatobiliary disorders) | 13 | 13 — According to investigators, the causal relationship with the study drug / standard therapy was estimated as "unrelated" in 69.2% /61.5%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT04542694/Prot_SAP_000.pdf